CLINICAL TRIAL: NCT05352373
Title: The Role of Dietary Calcium for the Treatment of Osteopenia in Girls With Rett Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Kathleen J Motil, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-19205
Record Dates: First submitted 2022-04-15; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Rett Syndrome
Keywords: Low bone mass
MeSH Terms: conditions — Rett Syndrome | interventions — Calcium

STUDY DESIGN:
Intervention Model Description: randomized, double blind
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rett Active Supplement (Active Comparator): Females with clinical diagnosis of Rett syndrome treated orally daily with calcium carbonate, dose based on Dietary Reference Intake for age, for one year
  Interventions: Dietary Supplement: calcium
- Rett Placebo Supplement (Placebo Comparator): Females with clinical diagnosis of Rett syndrome treated orally daily with sodium bicarbonate, dose based on equivalent weight for active supplement for age, for one year
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: calcium — calcium carbonate
  Arms: Rett Active Supplement
Dietary Supplement: placebo — sodium bicarbonate
  Arms: Rett Placebo Supplement

SUMMARY:
Randomized, placebo-controlled trial of oral calcium supplementation for osteopenia in girls and women with Rett syndrome

DETAILED DESCRIPTION:
Objective: The investigators conducted a randomized, double-blind, placebo-controlled trial to determine the safety and efficacy of oral calcium supplementation for the treatment of bone mineral deficits in individuals with Rett syndrome (RTT).

Methods: The investigators measured total body bone mineral content (BMC) and bone mineral density (BMD) by dual-energy x-ray absorptiometry and biomarkers of bone turnover by clinical laboratory techniques before and one year after oral calcium or placebo supplementation in 32 pre- and post-pubertal girls and young women with RTT. The calcium supplement was calculated to provide a twofold increase in the recommended dietary allowance of calcium for age.

ELIGIBILITY:
Inclusion Criteria

* clinical diagnosis of Rett syndrome

Exclusion Criteria

* parathyroid disease
* renal disease

Ages: 5 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral content (BMC) | change from baseline to 1 year thereafter
  Bone mineral content (z-score) measured by dual-energy x-ray absorptiometry
Bone mineral density (BMD) | change from baseline to 1 year thereafter
  Bone mineral density (z-score) measured by dual-energy x-ray absorptiometry

SECONDARY OUTCOMES:
Osteocalcin | change from baseline to 1 year thereafter
  Serum Osteocalcin (ng/ml)
Bone alkaline phosphatase | change from baseline to 1 year thereafter
  Serum Bone alkaline phosphatase (mcg/ml)
C-telopeptide | change from baseline to 1 year thereafter
  Serum C-telopeptide (pg/ml)
Calcium/creatinine ratio | change from baseline to 1 year thereafter
  Urinary calcium/creatinine ratio (mg/g)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen J Motil, MD, PHD, Principal Investigator — Baylor College of Medicine